CLINICAL TRIAL: NCT06633068
Title: The Analgesic Efficacy of Perineural Nalbuphine as an Adjuvant to Bupivacaine in Ultrasound Guided Superficial Cervical Plexus Nerve Block for Thyroid Surgeries. A Double Blinded Randomized Controlled Trial.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Yahia El Sayed Kamel, Lecturer of anesthesiology and surgical ICU and pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Nerve blocks
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Intra and Postoperative Pain Management

STUDY DESIGN:
Intervention Model Description: A double blinded randomized controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: • Patients will be randomized using a computer-generated randomization list. Random group assigned will be enclosed in a sealed envelope to ensure concealment of allocation sequence. The sealed envelope will be opened by an anaesthesiologist who will not be involved in the study to prepare the drug solution according to randomization. The anaesthesiologist performing the block and observing the patient will be blinded to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (C) control group (Placebo Comparator): Patients will receive bilateral superficial cervical plexus block with 28 ml bupivacine 0.25% mixed with 2 ml saline 0.9%, to a volume of 30 ml, 15 ml on each side of the neck before induction of general anaesthesia.
  Interventions: Drug: Adding perineural Nalbuphine to Bupivacaine in superficial cervical nerve block
- Group (N) Perineural Nalbuphine (Active Comparator): Patients will receive bilateral superficial cervical plexus block with 28 ml Bupivacaine 0.25% mixed with 10 mg nalbuphine in saline 0.9% to a volume of 30 ml, 15 ml on each side of the neck before induction of general anaesthesia.
  Interventions: Drug: Adding perineural Nalbuphine to Bupivacaine in superficial cervical nerve block

INTERVENTIONS:
Drug: Adding perineural Nalbuphine to Bupivacaine in superficial cervical nerve block — Adding nalbuphine as an adjuvant to bupivacaine in superficial cervical plexus block during thyroid surgeries

SUMMARY:
This study aiming to evaluate the analgesic effect of adding nalbuphine as an adjuvant to bupivacaine in superficial cervical plexus block during thyroid surgeries regarding first rescue analgesia in the first twenty-four hours postoperative, VAS score after extubation and complications such as postoperative nausea, vomiting and respiratory depression.

DETAILED DESCRIPTION:
Thyroidectomy is a common and painful procedure demanding analgesia. Patients may experience discomfort in swallowing, burning sensation in the throat, nausea, and vomiting, which are all caused by the surgical procedures or general anaesthesia. Thyroid surgeries induce brief postoperative pain caused by several mechanisms. One of the mechinsims of this Post-operative pain, believed to be due to the interruption of the rich nerve supply present in the neck.

A lot of drugs have been used to decrease this postoperative pain such as non-steroidal anti inflammatory drugs , opioids or regional blocks. Traditionally, opioids have been the mainstay of postoperative analgesia, specifically at thyroid and parathyroid surgical centers, where narcotic analgesics make up the major component of their postoperative pain control regimens. However, the use of opioids has been linked to an increased risk of postoperative complications that include ventilatory depression, sedation, postoperative nausea and vomiting (PONV), pruritis, difficulty of voiding, ileus and surgical site infections which can in turn contribute to delayed hospital discharge. Further acute and chronic opioids can have significant effects on the endocrine system. Longer-term use of opioids may lead to dependence and substance abuse disorder.

The skin overlying the neck, ear, angle of the mandible, shoulder, and clavicle is supplied by the superficial cervical plexus (SCP), which is a sensory neural plexus formed from the ventral rami of the first four cervical nerves (C1-C4). It emerges behind the posterior border of sternomastoid muscle.

Bilateral superficial cervical plexus block (SCPB) has shown good intraoperative and postoperative analgesia in upper neck surgeries especially in thyroidectomies, this regional block can be facilitated by using ultrasound guided technique as it provides good visualisation of the anatomical structures and decreases the complications.

There has always been a search for ideal adjuvants in peripheral nerve blocks which prolong the duration of analgesia with lesser adverse effects, Recently, nalbuphine was studied frequently as an adjuvant to local anesthetics in spinal and epidural and the results of all studies concluded that nalbuphine is effective when used as an adjuvant to local anaesthetics in spinal and epidural as it significantly prolongs the block duration.

The mechanism of perineural nalbuphine has not been clearly identified till now, previous studies demonstrated underlying mechanism could be interpreted that inflammatory response increases the synthesis of opioid receptors in the dorsal root ganglion neurons and enhances axonal transport and accumulation of opioid receptors in the sensory nerve endings in the inflamed tissue. Moreover, nalbuphine is an opioid receptors antagonist that allows for the peripheral analgesic effects of opioids in addition to the analgesic effect of its systemic absorption.

However, nalbuphine has not been studied extensively as an additive for peripheral nerve blocks as there was a minor research about it as an adjuvant to bupivacaine in brachial plexus block for upper limb surgeries and it showed that it prolongs the duration of sensory and motor blockades and reduces the requirement of analgesics in postoperative period. The superficial cervical block is a sensory block carrying sensory nerve fibers only with different axonal chemistry .

To our knowledge, no study till date compared the analgesic effect of perineural nalbuphine as an adjuvant to the superficial cervical block.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 to 60 years old of both sexes undergoing elective thyroid surgery.
* ASA I and II.

Exclusion Criteria:

* Patient refusal.
* Hypersensitivity or contraindication to nalbuphine or bupivacaine.
* Pregnancy or lactating mothers.
* Hepatic, cardiac or renal diseases.
* Bleeding disorders.
* Severe neurological or psychological disorders.
* Goitres with retrosternal extension.
* Any anatomical disruption in the neck (ex: metastatic lymph nodes).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
time to first rescue analgesia (will be given to VAS score > 4) following surgery in the first 24 hours. | First 24 hours postoperative
  defined as the time interval between the end of surgery and the first request to postoperative Nalbuphine

SECONDARY OUTCOMES:
Intraoperative hemodynamics | every 10 minutes until the end of the surgery
  mean arterial blood pressure
VAS score after extubation | at 0,2,6,12,18 and 24 hours after completion of surgery.
  Visual Analogue Scale (VAS) measures pain intensity.
Total amount of nalbuphine administrated to the patient 24 hours postoperative. | Every one hour postoperative for 24 hours
  As analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M Zayed, Assistant professor, Study Director — Cairo University; Amany Eissa, Doctorate, Study Director — Cairo University; Omnia Y Kamel, Doctorate degree, Study Director — Cairo University
Locations (1):
- Kasr Alainy Teaching Hospitals, Giza, الجيزة, Egypt